CLINICAL TRIAL: NCT02043704
Title: The Effect of Intravenous Acetaminophen on Post-operative Pain and Narcotic Consumption in Vaginal Reconstructive Surgery Patients: A Randomized Controlled Trial
Brief Title: RCT (Randomized Controlled Trial) of IV Acetaminophen for Post Operative Vaginal Reconstruction Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 13072
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Results first posted 2018-03-14 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-02

CONDITIONS: Post Operative Pain
Keywords: IV Acetaminophen; Vaginal Reconstruction; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV Acetaminophen (Experimental): Subjects will receive a 1000mg dose of IV acetaminophen in 100mL solution every 6 hours for 24 hours. The first dose will be administered prior to anesthesia induction, approximately 30 minutes before skin incision. A total of 4 doses will be given.
  Interventions: Drug: IV Acetaminophen
- Saline (Placebo Comparator): Subjects will receive a 100mL dose of IV saline every 6 hours for 24 hours. The first dose will be administered prior to anesthesia induction, approximately 30 minutes before skin incision. A total of 4 doses will be given.
  Interventions: Drug: IV Acetaminophen

INTERVENTIONS:
Drug: IV Acetaminophen — Details covered in arm description.
  Other Names: Ofirmev

SUMMARY:
This randomized controlled trial will evaluate the effects of perioperative intravenous (IV) acetaminophen on postoperative narcotic consumption and pain scores in subjects undergoing vaginal reconstructive surgery. One hundred subjects will be randomly assigned to receive either IV acetaminophen or IV placebo. Those in the IV acetaminophen group will receive 1000mg IV every 6 hours for 24 hours beginning prior to anesthesia induction. The control group will receive placebo saline infusions at the same time intervals. All subjects will receive as needed (prn) IV narcotic for additional pain relief. Visual analog scales (VAS) regarding pain will be evaluated at 18 and 24 hours postoperative and immediately prior to discharge. We will also collect total IV narcotic consumption. We hypothesize that subjects receiving IV acetaminophen will have lower VAS scores and decreased total narcotic consumption in comparison to the control group.

DETAILED DESCRIPTION:
see brief summary

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 70 years
* Patients of the Division of Urogynecology at Good Samaritan and Bethesda North Hospitals in Cincinnati, Ohio
* Scheduled to undergo major vaginal reconstruction
* Must undergo total vaginal hysterectomy, anterior repair, posterior repair, enterocele repair, and intraperitoneal vault suspension. The addition of suburethral sling is not a cause for exclusion.

Exclusion Criteria:

* Allergy to acetaminophen
* Liver disease (chronic or active)
* Chronic alcohol use (>1 drink/day)
* Bleeding diathesis
* Renal disease
* Opiate dependent or daily use
* History of chronic pain
* Mental or cognitive disorder preventing patient to accurately verbalize pain levels
* Undergoing abdominal or laparoscopic procedures at the time of surgery
* Allergy to hydromorphone
* Surgery is not performed under general anesthesia

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catrina Crisp, MD, MSc, Principal Investigator — TriHealth Inc.
Locations (1):
- TriHealth - Good Samaritan and Bethesda North Hospitals, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crisp CC, Khan M, Lambers DL, Westermann LB, Mazloomdoost DM, Yeung JJ, Kleeman SD, Pauls RN. The Effect of Intravenous Acetaminophen on Postoperative Pain and Narcotic Consumption After Vaginal Reconstructive Surgery: A Double-Blind Randomized Placebo-Controlled Trial. Female Pelvic Med Reconstr Surg. 2017 Mar/Apr;23(2):80-85. doi: 10.1097/SPV.0000000000000347. PMID 28230615

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IV Acetaminophen | Saline
Started | 50 | 50
Completed | 47 | 43
Not Completed | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Acetaminophen | Saline | Total
Number analyzed (Participants) | 47 | 43 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (12.8) | 59.4 (11.4) | 58.3 (12.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 43 | 90
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 47 | 43 | 90
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 47 | 43 | 90

OUTCOME MEASURES:

1. Primary Outcome: Pain While Active - 18 hr
Description: Post operative pain will be assessed 18 hours after surgery. Pain will be self reported by patients using a 0-100 mm visual analog scale (VAS) with 0 indicating no pain and 100 indicating the worst pain imaginable. A pain score will be collected for pain while active.
Time Frame: 18 hours
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | IV Acetaminophen | Saline
Number analyzed (Participants) | 47 | 43
mm | 42.0 [27.5 to 61] | 50.0 [28.5 to 71.5]
Statistical Analysis 1: Comparison: IV Acetaminophen vs Saline; The comparison was analyzed using the Mann-Whitney U test; Test type: Equivalence — The null hypothesis is that there is no difference in the pain scores between the groups; p = 0.328, Wilcoxon (Mann-Whitney) — The p-value was not adjusted for multiple comparisons; There were no adjustments

2. Primary Outcome: Total Amount of Narcotic Consumption in the First 24 Hours Post Surgery
Description: Hydromorphone will be administered for breakthrough pain. The total amount consumed in the first 24 hours post surgery will be recorded.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: mgs
Arm/Group | IV Acetaminophen | Saline
Number analyzed (Participants) | 47 | 43
mgs | 13 [6.67 to 26.68] | 15 [5 to 26.67]

3. Secondary Outcome: Narcotic Associated Side Effects
Description: The incidence of known narcotic associated side effects will be recorded for nausea/vomiting.
Time Frame: 24 hours
Population: Count reported for nausea/vomiting.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen | Saline
Number analyzed (Participants) | 47 | 43
Participants | 27 | 22

4. Secondary Outcome: Time to First Rescue Narcotic
Description: The time from the end of surgery to the time any IV narcotic is given.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | IV Acetaminophen | Saline
Number analyzed (Participants) | 47 | 43
minutes | 27 [18 to 64] | 41 [22 to 67]

5. Secondary Outcome: Narcotic Associated Side Effects
Description: The incidence of known narcotic associated side effects will be recorded for itching.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen | Saline
Number analyzed (Participants) | 47 | 43
Participants | 11 | 5

6. Secondary Outcome: Narcotic Associated Side Effects
Description: The incidence of known narcotic associated side effects will be recorded for headache.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen | Saline
Number analyzed (Participants) | 47 | 43
Participants | 6 | 3

7. Secondary Outcome: Narcotic Associated Side Effects
Description: The incidence of known narcotic associated side effects will be recorded for insomnia.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen | Saline
Number analyzed (Participants) | 47 | 43
Participants | 8 | 2

8. Secondary Outcome: Narcotic Associated Side Effects
Description: The incidence of known narcotic associated side effects will be recorded for rash/hives.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen | Saline
Number analyzed (Participants) | 47 | 43
Participants | 0 | 0

9. Secondary Outcome: Narcotic Associated Side Effects
Description: The incidence of known narcotic associated side effects will be recorded for shortness of breath.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen | Saline
Number analyzed (Participants) | 47 | 43
Participants | 4 | 0

10. Secondary Outcome: Narcotic Associated Side Effects
Description: The incidence of known narcotic associated side effects will be recorded for respiratory depression.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen | Saline
Number analyzed (Participants) | 47 | 43
Participants | 0 | 0

11. Secondary Outcome: Narcotic Associated Side Effects
Description: The incidence of known narcotic associated side effects will be recorded for urinary retention.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen | Saline
Number analyzed (Participants) | 47 | 43
Participants | 29 | 20

12. Secondary Outcome: Time to Ambulation
Description: Length of time from the end of surgery to the time of ambulation.
Time Frame: 1800 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | IV Acetaminophen | Saline
Number analyzed (Participants) | 47 | 43
minutes | 1295 [1108 to 1462] | 1252 [778 to 1459]

13. Other Pre Specified Outcome: Time to First Flatus/Bowel Movement
Description: Length of time from the end of surgery to the time of first flatus or bowel movement.
Time Frame: 9000 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | IV Acetaminophen | Saline
Number analyzed (Participants) | 47 | 43
minutes | 3977 [1437 to 5564] | 1899 [1275 to 4580]

ADVERSE EVENTS:
Arm/Group | IV Acetaminophen | Saline
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes